CLINICAL TRIAL: NCT04381858
Title: Efficacy and Safety of Convalescent Plasma vs Human Immunoglobulin for the Treatment of COVID-19 Pneumonia: A Randomized Controlled Trial
Brief Title: Convalescent Plasma vs Human Immunoglobulin to Treat COVID-19 Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A-10
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-05

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe pneumonia due to COVID-19 (Experimental): Patients who are admitted to Hospital Centers with a positive RT-qPCR SARS-CoV-2 test or a CT scan compatible with a diagnosis of COVID-19 pneumonia, in addition to one of the following two criteria:
  1. Severe respiratory failure [respiratory rate> 25 - <35 x minute, oxygen saturation ≤ 90% with reservoir mask (FiO2 = 100%)]
  2. Requiring invasive mechanical ventilation.
  Interventions: Drug: Plasma from COVID-19 convalescent patient
- Severe pnemonia due to COVID-19 (Active Comparator): Patients who are admitted to Hospital Centers with a positive RT-qPCR SARS-CoV-2 test or a CT scan compatible with a diagnosis of COVID-19 pneumonia, in addition to one of the following two criteria:
  1. Severe respiratory failure [respiratory rate> 25 - <35 x minute, oxygen saturation ≤ 90% with reservoir mask (FiO2 = 100%)]
  2. Requiring invasive mechanical ventilation.
  Interventions: Drug: Human immunoglobulin

INTERVENTIONS:
Drug: Plasma from COVID-19 convalescent patient — Infusion of 400 ml (2 units) of plasma.
  Plasma donated from convalescent patients will be extracted in strict compliance with the following criteria:
  * History of a clinical event with symptoms attributed to COVID-19 and a positive PCR test for COVID-19
  * Further confirmation of a negative PCR test for COVID-19
  * In order to be eligible plasma donors must complete at least 14 days after the last negative PCR in the absence of any symptom attributable to COVID-19 infection
  * IgG antibodies for COVID-19 must be confirmed POSITIVE when a qualitative assay is being used
  * When quantification of IgG antibodies for COVID-19 is available a title > 1: 640 will be required for inclusion.
  * Apheresis will be used as the only method for plasma extraction.
  Arms: Severe pneumonia due to COVID-19
Drug: Human immunoglobulin — Human immunoglobulin 0.3 gr/kg/day (5 doses)
  Arms: Severe pnemonia due to COVID-19

SUMMARY:
Background: On December 2019, a new human coronavirus infection (COVID-19) was detected in China. Its infectivity and virulence characteristics caused a rapid spread, being declared pandemic on March 2020. The mortality attributed to the infection ranges between 3 and 10%. Main risk factors are age, male sex, and chronic degenerative comorbidities. Due to the absence of therapeutic options, potential alternatives such as human immunoglobulin or plasma from convalescent patients have been administered. Due to the severity of the disease and the associated mortality, it is urgent to find therapeutic alternatives.

Objective: To assess the safety and efficacy of the administration of Convalescent plasma vs human immunoglobulin in critically ill patients with COVID-19 infection.

Material and methods: Randomized Controlled trial of patients diagnosed with respiratory infection by COVID-19, with severe respiratory failure without indication of mechanical ventilation, or those who due to their severity are intubated upon admission. Randomization will be performed 2:1 to receive plasma from convalescent patients or human immunoglobulin.

Outcomes: The primary outcome will be time to discharge from hospital for improvement. The safety outcomes will be: Kirby index (PaO2/FiO2) evolution and dead.

DETAILED DESCRIPTION:
I. Background:

In late December 2019, the health authorities of the Popular Republic of China reported several cases of pneumonia of unknown origin in Wuhan City, Hubei Province, China. On December 31, 2019, the Chinese Center for Disease Control and Prevention began etiological and epidemiological research on this disease. Three samples of bronchoalveolar lavage were taken from patients from the Jinyintan hospital in Wuhan and through various processes they came to identify a new coronavirus that they initially called on January 7, 2020 as: 2019-nCoV. On January 2020, the World Health Organization (WHO) made the first recommendations on the epidemiological surveillance of this new coronavirus.

On January 22, 2020, the first session of the Emergencies Committee was convened by WHO in Geneva, Switzerland and on January 30 a Public Health Emergency of International Importance (ESPII) was declared.

On February 11, the International Committee on Virus Taxonomy named this new coronavirus as SARS-CoV-2 and responds to "Severe Acute Respiratory Syndrome Coronavirus 2 "(Severe Acute Respiratory Syndrome CoronaVirus 2), the WHO proposes that same day to call the disease caused by SARS-CoV-2 as COVID-19.

The first case reported in Latin America was in Brazil on February 26 and on the 28th of the same month, Mexico communicates its first confirmed case of the new coronavirus in a 35-year-old patient from a trip to Italy.

Given the alarming levels of spread and severity of COVID-19, on March 11, WHO Director-General Tedros Adhanom Ghebreyesus declares the SARS-CoV-2.5 outbreak as a pandemic. A high percentage of patients especially over 50 y with comorbidities require hospitalization and intensive care. Mortality of patients with invasive mechanical intubation has been reported up to 61% .

At this time, there are no treatment that has shown clinical efficacy, so the plasma from convalescent patients and human immunoglobulin (IVIG) have been proposed as alternatives.

Human immunoglobulin:

There are no controlled studies with the use of IVIG for the treatment of COVID-19 infection. In observational reports it was found in three patients with early forms in patients hospitalized for pneumonia secondary to COVID-19, treated with IVIG at a dose of 0.3 - 0.5 gr / kg. All three patients showed clinical improvement, so this study justified the start of a clinical trial.

An observational experience with important limitations in its report, describes the experience with 58 patients with severe pneumonia who found differences in mortality at 28 days when they divided the groups according to the IVIG administration time (48 hours), emphasizing the importance of early application.

In similar situations historically diverse scenarios have been found where IVIG has been administered with apparent success. However, there are no clinical trials supporting its use.

Convalescent patient plasma:

The use of plasma from convalescent patients for the treatment of severe infection by COVID19 has been considered as a first-line therapeutic option since the start of the pandemic. The seroconversion of the patients during the first months of the outbreak was unknown, being an obstacle to recommend this type of treatment. Very recently, the serological behavior of 285 patients was published; 100% of the patients have detected antibodies 19 days after detection of the virus.

The experiences reported so far are only case series without simultaneous comparative groups. Viral clearance has been effective, in all included patients in a small series of 6 patients. This viral clearance was not accompanied by mortality benefits, the authors suggesting that it was probably due to the late administration of plasma.

Data supporting the use of convalescent plasma for severe acute respiratory syndrome (SARS) are limited to case reports and case series. Use in case series for severe infections due to MERS, Ebola and influenza have reported clinical improvement, although none of the studies were conducted comparatively.

Risks associated with plasma transfusion include TRALI, transfusion-associated circulatory overload, and allergic transfusion reactions. Rare complications include transmission of infectious diseases and alloimmunization of red blood cells.

Clinical trials are underway to evaluate both convalescent plasma and IVIG from SARS-CoV-2 for the treatment of COVID-19.

The FDA has approved a national expanded access program for the use of convalescent plasma for the treatment of patients with COVID-19. Physicians can refer to the National Convalescent Plasma Project COVID-19 website for more information. People who have fully recovered from COVID-19 for at least two weeks and are interested in donating plasma can contact their local blood donor or plasma collection center or consult the American Red Cross website.

The national transfusion center in Mexico has published guidelines for the use of serum from convalescent patients.

II. Definition of the problem:

COVID-19 infection has had a high rate of spread. In patients with comorbidities and over 50 years, the infection has presented the highest rate of respiratory deterioration and the requirement for invasive mechanical ventilation. Due to the absence of specific treatment, various alternatives have been explored. In critically ill patients, the administration of human immunoglobulin and plasma from convalescent patients have emerged as potential rescue therapies. The proposed treatments have an adequate margin of safety due to routine clinical use in other settings. Due to this, in conjunction with the urgent need to seek therapeutic alternatives, controlled studies are required without assuming efficacy.

III. Justification COVID-19 infection has collapsed health systems in almost all the countries due to the large number of patients requiring respiratory assistance.

There is no standard treatment for the management of this infection and the focus has been on the already known life support and management of Adult Respiratory Distress Syndrome in critically ill patients.

The treatments used empirically have an adequate safety profile due to the experience in other clinical settings.

The use of these empirical alternatives should be based on clinical trials since efficacy and safety should not be assumed in the group of patients with COVID-19.

The Miguel Hidalgo Centennial Hospital has been designated as a hospitalization center for COVID-19 patients who do not have Social Security in the state of Aguascalientes.

IV. Hypothesis

In patients with COVID19 infection with severe respiratory failure or requiring invasive mechanical ventilation, plasma treatment of convalescent patients will be superior to immunoglobulin, with a shorter hospital stay and a lower rate of complications: deterioration of the oxygenation index or death.

V. General objectives.

To assess the safety and efficacy of plasma administration of convalescent patients or immunoglobulin in patients with severe COVID-19 infection with severe respiratory failure or requiring mechanical ventilation.

Assess viral clearance time using PCR

VI. Methodology

Randomized controlled trial, Included patients will be randomized (2:1) to receive one of two maneuvers:

Group 1: Plasma donated from convalescent patients will be extracted in strict compliance with the following criteria:

* History of a clinical event with symptoms attributed to COVID-19 and a positive PCR test for COVID-19
* Further confirmation of a negative PCR test for COVID-19
* In order to be eligible plasma donors must complete at least 14 days after the last negative PCR in the absence of any symptom attributable to COVID-19 infection
* IgG antibodies for COVID-19 must be confirmed POSITIVE when a qualitative assay is being used
* When quantification of IgG antibodies for COVID-19 is available a title > 1: 640 will be required for inclusion.
* Apheresis will be used as the only method for plasma extraction. Infusion of 400 ml of Plasma will be infused

Group 2: Human immunoglobulin 0.3 gr / kg (5 doses)

VII. Definition of the variables:

Days of hospitalization: Days from admission as a suspected case of COVID with hospitalization criteria until discharge.

Hospital discharge criteria: negative PCR for COVID-19, oxygen saturation in ambient air > 90%, absence of fever and dyspnea.

Oxygen supplementation requirement: This is based on the modality and FiO2 necessary to maintain a saturation of 90% of ambient air without respiratory distress.

Respiratory distress syndrome: Respiratory rate greater than 25 x minute and use of accessory muscles.

Respiratory failure: Saturation to ambient air below 90% or PO2 below 60 mmHg. Septic Shock: Requirement of vasoactive amines to maintain mean arterial pressure above 65 mmHg, in a patient previously with adequate water resuscitation.

SOFA: Organic failure scale that includes: PaO2 / FiO2 ratio, platelet count, bilirubin, blood pressure, Glasgow scale and kidney function.

APACHE 2: Morbidity scale in intensive care. PaO2 / FiO2 Index: Ratio of oxygen pressure to inspired fraction of oxygen RT-qPCR SARS-CoV-2: Quantitative measurement by RT-PCR method usually performed on blood. It will be evaluated as a start for diagnosis and then a test will be repeated on days 5, 14 and 21 to assess viral clearance.

Inflammatory markers: Laboratory studies used as markers of disease severity, consist of procalcitonin, C-reactive protein, lactate dehydrogenase, blood cytometry, dimer-D, ferritin.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to Hospital Centers with a positive RT-qPCR SARS-CoV-2 test or a CT scan compatible with a diagnosis of COVID-19 pneumonia, in addition to one of the following two criteria:

  1. Severe respiratory failure [respiratory rate> 25 - <35 x minute, oxygen saturation ≤ 90% with reservoir mask (FiO2 = 100%)]
  2. Requiring invasive mechanical ventilation.

Exclusion Criteria:

* Patients with a viral infection other than COVID-19

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Mean hospitalization time | Through study completion, an average of 3 months
  Mean days from admission as a suspected case of COVID with hospitalization criteria until discharge
Mean Oxigenation index evolution | Through study completion, an average of 3 months
  Mean of delta of oxigenation index (PaO2/FiO2)
Rate of severe ARDS | Through study completion, an average of 3 months
  Rate of patients with evolution to severe ARDS (PaO2/FiO2 < 100)
Rate and time to dead | Through study completion, an average of 3 months
  Rate of Dead caused by COVID-19 related complications and time to dead caused by COVID-19 complication
Mean time with invasive mechanical ventilation | Through study completion, an average of 3 months
  Mean time with invasive mechanical ventilation

SECONDARY OUTCOMES:
Time to Viral PCR Negativization | Through study completion, an average of 3 months.
  Time to negativization of RT-qPCR SARS-CoV-2 test.

CONTACTS AND LOCATIONS:
Locations (1):
- Centenario Hospital Miguel Hidalgo, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Lv DF, Ying QM, Weng YS, Shen CB, Chu JG, Kong JP, Sun DH, Gao X, Weng XB, Chen XQ. Dynamic change process of target genes by RT-PCR testing of SARS-Cov-2 during the course of a Coronavirus Disease 2019 patient. Clin Chim Acta. 2020 Jul;506:172-175. doi: 10.1016/j.cca.2020.03.032. Epub 2020 Mar 27. PMID 32229107
- [Background] Munster VJ, Koopmans M, van Doremalen N, van Riel D, de Wit E. A Novel Coronavirus Emerging in China - Key Questions for Impact Assessment. N Engl J Med. 2020 Feb 20;382(8):692-694. doi: 10.1056/NEJMp2000929. Epub 2020 Jan 24. No abstract available. PMID 31978293
- [Background] Correction to Lancet Infect Dis 2020; published online March 11, https://doi.org/10.1016/ S1473-3099(20)30144-4. Lancet Infect Dis. 2020 May;20(5):e79. doi: 10.1016/S1473-3099(20)30251-6. Epub 2020 Mar 25. No abstract available. PMID 32220652
- [Background] Cao W, Liu X, Bai T, Fan H, Hong K, Song H, Han Y, Lin L, Ruan L, Li T. High-Dose Intravenous Immunoglobulin as a Therapeutic Option for Deteriorating Patients With Coronavirus Disease 2019. Open Forum Infect Dis. 2020 Mar 21;7(3):ofaa102. doi: 10.1093/ofid/ofaa102. eCollection 2020 Mar. PMID 32258207
- [Background] Xie Y, Cao S, Dong H, Li Q, Chen E, Zhang W, Yang L, Fu S, Wang R. Effect of regular intravenous immunoglobulin therapy on prognosis of severe pneumonia in patients with COVID-19. J Infect. 2020 Aug;81(2):318-356. doi: 10.1016/j.jinf.2020.03.044. Epub 2020 Apr 10. No abstract available. PMID 32283154
- [Background] Wang JT, Sheng WH, Fang CT, Chen YC, Wang JL, Yu CJ, Chang SC, Yang PC. Clinical manifestations, laboratory findings, and treatment outcomes of SARS patients. Emerg Infect Dis. 2004 May;10(5):818-24. doi: 10.3201/eid1005.030640. PMID 15200814
- [Background] Bloch EM, Shoham S, Casadevall A, Sachais BS, Shaz B, Winters JL, van Buskirk C, Grossman BJ, Joyner M, Henderson JP, Pekosz A, Lau B, Wesolowski A, Katz L, Shan H, Auwaerter PG, Thomas D, Sullivan DJ, Paneth N, Gehrie E, Spitalnik S, Hod EA, Pollack L, Nicholson WT, Pirofski LA, Bailey JA, Tobian AA. Deployment of convalescent plasma for the prevention and treatment of COVID-19. J Clin Invest. 2020 Jun 1;130(6):2757-2765. doi: 10.1172/JCI138745. PMID 32254064
- [Background] Long QX, Liu BZ, Deng HJ, Wu GC, Deng K, Chen YK, Liao P, Qiu JF, Lin Y, Cai XF, Wang DQ, Hu Y, Ren JH, Tang N, Xu YY, Yu LH, Mo Z, Gong F, Zhang XL, Tian WG, Hu L, Zhang XX, Xiang JL, Du HX, Liu HW, Lang CH, Luo XH, Wu SB, Cui XP, Zhou Z, Zhu MM, Wang J, Xue CJ, Li XF, Wang L, Li ZJ, Wang K, Niu CC, Yang QJ, Tang XJ, Zhang Y, Liu XM, Li JJ, Zhang DC, Zhang F, Liu P, Yuan J, Li Q, Hu JL, Chen J, Huang AL. Antibody responses to SARS-CoV-2 in patients with COVID-19. Nat Med. 2020 Jun;26(6):845-848. doi: 10.1038/s41591-020-0897-1. Epub 2020 Apr 29. PMID 32350462
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Zeng QL, Yu ZJ, Gou JJ, Li GM, Ma SH, Zhang GF, Xu JH, Lin WB, Cui GL, Zhang MM, Li C, Wang ZS, Zhang ZH, Liu ZS. Effect of Convalescent Plasma Therapy on Viral Shedding and Survival in Patients With Coronavirus Disease 2019. J Infect Dis. 2020 Jun 16;222(1):38-43. doi: 10.1093/infdis/jiaa228. PMID 32348485
- [Background] Chun S, Chung CR, Ha YE, Han TH, Ki CS, Kang ES, Park JK, Peck KR, Cho D. Possible Transfusion-Related Acute Lung Injury Following Convalescent Plasma Transfusion in a Patient With Middle East Respiratory Syndrome. Ann Lab Med. 2016 Jul;36(4):393-5. doi: 10.3343/alm.2016.36.4.393. No abstract available. PMID 27139619
- [Background] Burnouf T, Radosevich M. Treatment of severe acute respiratory syndrome with convalescent plasma. Hong Kong Med J. 2003 Aug;9(4):309; author reply 310. No abstract available. PMID 12904626
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Kong L. Severe acute respiratory syndrome (SARS). Transfus Apher Sci. 2003 Aug;29(1):101. doi: 10.1016/s1473-0502(03)00109-5. No abstract available. PMID 12952008
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Beigel JH, Tebas P, Elie-Turenne MC, Bajwa E, Bell TE, Cairns CB, Shoham S, Deville JG, Feucht E, Feinberg J, Luke T, Raviprakash K, Danko J, O'Neil D, Metcalf JA, King K, Burgess TH, Aga E, Lane HC, Hughes MD, Davey RT; IRC002 Study Team. Immune plasma for the treatment of severe influenza: an open-label, multicentre, phase 2 randomised study. Lancet Respir Med. 2017 Jun;5(6):500-511. doi: 10.1016/S2213-2600(17)30174-1. Epub 2017 May 15. PMID 28522352
- [Background] Narick C, Triulzi DJ, Yazer MH. Transfusion-associated circulatory overload after plasma transfusion. Transfusion. 2012 Jan;52(1):160-5. doi: 10.1111/j.1537-2995.2011.03247.x. Epub 2011 Jul 18. PMID 21762464
- [Background] Sheridan C. Convalescent serum lines up as first-choice treatment for coronavirus. Nat Biotechnol. 2020 Jun;38(6):655-658. doi: 10.1038/d41587-020-00011-1. No abstract available. PMID 32358594
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- See also: Statement on the second meeting of the International Health Regulations (2005) Emergency Committee regarding the outbreak of novel coronavirus 2019 (n-CoV) on 30 January 2020. — http://www.who.int/news-room/detail/30-01-2020-statement-on-the-second-meeting-of-the-international-health-regulations-(2005)-emergency-committee-regarding-the-outbreak-of-novel-coronavirus-(2019-ncov)
- See also: World Health Organization.Coronavirus disease (COVID-19) outbreak — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: The feasibility of convalescent plasma therapy in severe COVID-19 patients: a pilot study — https://www.medrxiv.org/content/10.1101/2020.03.16.20036145v1
- See also: Registration format of research protocols related to the therapeutic use of plasma from convalescent donors of COVID-19 secondary to infection by SARS-CoV-2 - CNTS. National Center for Blood Transfusion — http://www.gob.mx/cnts